CLINICAL TRIAL: NCT02408874
Title: Study to Assess the Impact of Inhaled Silver Nanoparticles on Lung Cell Immune Response
Brief Title: Inhaled Nanosilver Study
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150104; 15-E-0104
Record Dates: First submitted 2015-04-03; First posted 2015-04-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-11-20

CONDITIONS: Inflammatory Disease
Keywords: Nanoparticles; Inflammatory Response; Silver; Lung Function; Lung Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Nanosilver is tiny silver particles. Many products contain nanosilver, like antimicrobial cleaning supplies and antimicrobial fabrics. Some products also contain nanosilver in a solution that people inhale. The companies that make these products claim they can help boost the immune system.

Objective:

- To learn if inhaling nanosilver affects the lung s immune system. In addition, to see if nanosilver affects lung function and if it gets absorbed into the bloodstream after it is inhaled.

Eligibility:

- Healthy, non-smoking adults ages 18 60.

Design:

* Participants will be pre-screened by phone.
* Participants will then be screened with a medical history and physical exam. They will give blood and urine samples.
* Participants will have lung function tests. They will breathe into a spirometer. It has a mouthpiece attached to a tube that is connected to a computer.
* Participants will have a methacholine challenge test. They will blow into a spirometer. Then they will inhale methacholine.
* Eligible participants will have 3 study visits over 2 5 weeks. At each visit, they will repeat some of the screening tests.
* At visit 1, participants will have a bronchoscopy. For this, an intravenous line is placed in an arm vein. Electrodes are placed on the chest. A tube is placed through the nose and into the airways. The airway is washed. A sample of cells is taken.
* At visit 2, participants will get the study treatment. They will inhale a nanosilver solution mist. They will have lung function tests before and after treatment.
* Participants will collect their urine from the time they get the treatment until they return to the clinic the next day.
* At visit 3, participants will turn in their urine. They will have another bronchoscopy.

DETAILED DESCRIPTION:
This is a single-center, single-arm pilot study to assess the impact of inhaled silver nanoparticles (nanosilver or nAg) on immune responses in the lung. Non-smoking, healthy adults (no lung or cardiovascular conditions), age 18-60 will be recruited to participate; pregnant or breastfeeding women will be excluded.

Potential participants will be prescreened by telephone and scheduled for a final eligibility visit that will include vital signs/anthropometry, medical/medication history review, physical exam, urine tests, blood draw, urine collection, and pulmonary function tests (PFTs; i.e., spirometry and methacholine challenge test). After eligibility is confirmed, the participant will be scheduled for a baseline visit, which includes vital signs/anthropometry, medical/medication history review, physical exam, blood draw, urine collection, and bronchoscopy (with lavage and brushing). Participants will return 14-40 days between the baseline visit and study treatment visit, which includes vital signs/anthropometry, blood draw, urine collection, spirometry, one-time administration of ionic silver via nebulizer, and instructions to collect urine for 24 hours. The next day after the study treatment visit, the participant will return for a visit that includes vital signs/anthropometry, blood draw, providing the 24-hour urine sample, spirometry, and bronchoscopy. During each bronchoscopy procedure, bronchoalveolar lavage (BAL) fluid and tissue from bronchial brushings will be collected from the participant to obtain alveolar macrophages and bronchial epithelial cells.

The primary objective of the study is to determine whether exposure to nanosilver alters the immune responses of lung cells. The primary laboratory analysis will determine whether exposure to nanosilver mediates a change from baseline in the response of bronchoscopy-derived, cultured macrophages or epithelial cells to challenge with a toll-like receptor (TLR) agonist. Additional analyses will assess changes in cytokine levels in BAL fluid, changes in the lung microbiome, silver penetration into the blood stream, silver excretion in the urine, and changes in PFT measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet all of the following criteria for enrollment:

1. Age 18 to 60 years (males and females)
2. Able to understand and provide written consent
3. Able to travel to the NIEHS CRU for required study visits
4. Able to present a valid government-issued form of identification for entry to the NIEHS campus
5. Able to fast for 6 hours prior to two visits where bronchoscopy occurs

EXCLUSION CRITERIA:

Participants meeting any of the following criteria at screening will not be eligible for enrollment:

1. Women who are pregnant or breastfeeding
2. Current smoker or significant second-hand smoke exposure (defined by urine cotinine >200 ng/mL at screening)
3. Body Mass Index (BMI) >35
4. Significant sources of exposure to silver that, in the investigator's opinion, will compromise the integrity of the study assessments (e.g., regular use of silver-containing dietary supplements, homeopathic remedies, or cleaning products)
5. FEV1 <80% predicted; or, positive methacholine test [i.e., provocative concentration of methacholine producing a 20% fall in FEV1 (PC20-FEV1) is reached at a solution of less than or equal to 4 mg/mL]
6. History of pulmonary or cardiovascular conditions, including the following comorbidities: chronic obstructive pulmonary disease, cystic fibrosis (CF), non-CF bronchiectasis, pulmonary fibrosis, sarcoidosis, pulmonary hypertension, unstable angina
7. Allergy or history of adverse reactions to metals
8. Any condition that, in the investigator's opinion, places the patient at undue risk for complications associated with required study procedures
9. Bleeding disorders
10. Facial deformity, major facial surgery
11. Allergy or history of adverse reactions to methacholine or lidocain (or other similar topical anesthetics)
12. Temperature >37.6 C, blood pressure <90/50 or >170/95 mmHg, or pulse rate <50 or >100 beats/minute (if in the investigator s clinical judgment, the exclusionary condition(s) may resolve, the candidate may be rescreened at a later date)
13. Body weight <50 kg (<110 lbs)
14. The following abnormal lab values on the screening blood work:

    * Platelet count <100,000/microliters
    * White blood cells count less than or equal to 1000/microliters
    * Absolute neutrophil count less than or equal to 500/microliters
    * Hematocrit <35% for both female and male
    * Hemoglobin less than or equal to 9 g/dL
    * Prothrombin Time (PT) / International Normalized Ratio (INR) greater than or equal to 1.3
    * Activated partial prothromboplastin time (aPTT) greater than or equal to 40 seconds
    * Serum creatinine greater than or equal to 1.4 mg/dL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-03; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of nanosilver exposure on ex vivo inflammatory response of bronchoscopy-derived cells (i.e. alveolar macrophage and epithelial cells) to challenge with a TLR agonist | 1 day post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)